CLINICAL TRIAL: NCT03720886
Title: Two-dose, Positive Drug Control, Multicentre, Randomized, Double-blind Study of Recombinant Human Parathyroid Hormone for Injection(rhPTH)(1-34) Once a Week to Treat Postmenopausal Osteoporosis Women for the Evaluation the Pharmacokinetics and Safety and to Explore Therapeutic Effects
Brief Title: G56W1 in Women With Postmenopausal Osteoporosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G56W1A201
Record Dates: First submitted 2018-10-14; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rhPTH（1-34） 28.2μg (Experimental): Participants received 28.2μg rhPTH（1-34）administered by subcutaneous injection once a week for 24 weeks.
  Interventions: Biological: rhPTH（1-34） 28.2μg
- rhPTH（1-34） 56.5μg (Experimental): Participants received 56.5μg rhPTH（1-34）administered by subcutaneous injection once a week for 24 weeks.
  Interventions: Biological: rhPTH（1-34） 56.5μg
- teriparatide acetate(Teribone™) (Active Comparator): Participants received 56.5μg teriparatide acetate(Teribone™) administered by subcutaneous injection once a week for 24 weeks.
  Interventions: Biological: teriparatide acetate(Teribone™)

INTERVENTIONS:
Biological: rhPTH（1-34） 28.2μg — Administered by subcutaneous injection
  Other Names: G56W1
  Arms: rhPTH（1-34） 28.2μg
Biological: rhPTH（1-34） 56.5μg — Administered by subcutaneous injection
  Other Names: G56W1
  Arms: rhPTH（1-34） 56.5μg
Biological: teriparatide acetate(Teribone™) — Administered by subcutaneous injection
  Arms: teriparatide acetate(Teribone™)

SUMMARY:
This study will assess the pharmacokinetics and safety and explore therapeutic effects with once-weekly recombinant human parathyroid hormone for injection ( 1-34 ) ( G56W1 ) in women with post-menopausal osteoporosis .The anticipated time on study treatment is 24 weeks, and the target sample size is 148 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Female, capable of self - motivation , 45 years old ≤ age ≤ 75 years old.
* Natural menopause for 3 years or more; or surgical menopause for 3 years or more (surgery needs to be performed after 40 years old), for women with surgical menopause, estradiol(E2)< 25 pg/ml and follicle stimulating hormone(FSH) > 40mIU/ml should be met.
* Weight ≥ 40kg , 18 ≤ body mass index(BMI)≤ 30 .
* Meets one of the following diagnostic criteria for osteoporosis, and ≥ 3 vertebral bodies of L1-4 can be measured by bone mineral density using the DXA method.

  1. Brittle fracture of the hip or vertebral body, and the bone density measurement T- score< -1.0.
  2. The T- score of the central axis bone mineral density or the 1/3 bone density of the distal radius of the tibia was ≤-2.5 measured by DXA .
  3. Bone density measurements were consistent with low bone mass ( -2.5 < T- value < -1.0 ) and combined with proximal humerus, pelvic or forearm distal brittle fractures.
* to participate in the trial and sign the informed consent form.

Exclusion Criteria:

* to have diseases affecting calcium or bone metabolism that are not effectively controlled, such as primary hyperparathyroidism or hyperthyroidism, Paget's bone disease, hypercalcemia, hypocalcemia, active urolithiasis.
* Secondary osteoporosis, such as osteomalacia, rheumatoid arthritis, gout, multiple myeloma, etc.
* Severe lumbar anatomical abnormalities which affecting DXA bone mineral density measurement, such as severe scoliosis.
* Patients who have been treated for anti-osteoporosis before random enrollment:

  1. Patients who received parathyroid hormone(PTH) therapy before random enrollment (including clinical trials of similar products).
  2. Patients who received bisphosphonate injection within 1 year prior to random enrollment or received bisphosphonate oral administration within 3 months for > 2 weeks prior to enrollment.
  3. Systemic treatment of androgen, estrogen, and selective estrogen receptor modulator(SERM) preparations within 3 months > 2 weeks prior to random enrollment.
  4. Three months before randomized to receive of heparin, warfarin, anticonvulsants (except benzodiazepines), digoxin accumulated for> 2 weeks.
  5. In the 3 months prior to random enrollment , received calcitonin, vitamin K preparation, active vitamin D3 preparation, oral or intravenous glucocorticoid treatment for > 4 weeks.
* Suffering from severe kidney disease, uncontrolled high blood pressure ( ≥150/100 mmHg ), symptomatic ischemic heart disease, cerebral infarction or obliterative atherosclerosis, malignancy, and other serious underlying diseases.
* Laboratory tests indicates abnormal, including any of the following indicators abnormalities (according to the normal range of each center, after consideration of the investigator with clinical considerations, such as caused by operational procedures, etc., after discussion with the sponsor, may allow retesting once) .

  1. Alkaline phosphatase(ALP)>1.5 times the upper limit of normal.
  2. Aspartate transaminase(AST) or alanine aminotransferase(ALT) or total bilirubin(TBIL) > 2.0 times the upper limit of normal.
  3. Glycated hemoglobin(HbA1c )≥ 7.0% .
  4. White blood cell(WBC)< 3.5×10^9 /L , Hb<100g/L or Plt<90×10^9 /L.
  5. Thyroid-stimulating hormone(TSH)<0.01 mIU/L (mU/L) or TSH>10 mIU/L (mU/L) .
  6. Parathyroid hormone(PTH)>1.5 times the upper limit of normal.
  7. Serum creatinine(SCr)>1.2 times the upper limit of normal.
  8. Serum total calcium(SCa)> normal upper limit.
* Subjects who had significant clinical significance including HIV , hepatitis B, hepatitis C, and syphilis ( hepatitis B virus carriers can be enrolled ) .
* Heavy Smoking (average of more than 10 / day) and / or alcohol addicted (converted to pure alcohol 30 ml / day or more) .
* Recent drug abuse or drug dependence evidence.
* Those who are allergic to test drugs / control drugs or biological products.
* Included in other interventional clinical trials within 3 months of the study.
* Been undergone radiation therapy for bones.
* Mental illness or any cause of cognitive impairment.
* Patients who were considered unsuitable for the study based on risk benefits by investigators.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
The percentage change in bone density of the lumbar spine ( L1-4 ) from baseline to 24 weeks after treatment | Baseline，week 24
  bone mineral density(BMD) measured by dual energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Evaluate the rate of change of Procollagen I N-terminal peptide(PINP),Serum cross-linked C-terminal telopeptide of type I collagen(s-CTX) ,Bone alkaline phosphatase(BALP) , and blood calcium from baseline | Baseline，week 24
  Central lab will be used
The percentage change of total hip bone density from baseline to 24 weeks after G56W1 treatment | Baseline，week 24
  BMD measured by DXA
Maximum plasma concentration (Cmax) | Baseline，week 1，week 4，week 12，week 24
  serum parathyroid hormone(PTH) will be tested for all pharmacokinetics parameters
Area under the plasma concentration versus time curve (AUC) | Baseline，week 1，week 4，week 12，week 24
  serum PTH will be tested for all pharmacokinetics parameters
Time to maximum plasma concentration（Tmax） | Baseline，week 1，week 4，week 12，week 24
  serum PTH will be tested for all pharmacokinetics parameters
Elimination half-life（t1/2） | Baseline，week 1，week 4，week 12，week 24
  serum PTH will be tested for all pharmacokinetics parameters

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, Prof., Principal Investigator — Peking Union Medical College
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital, Wanzhou, Chongqing Municipality
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - The West China Second UniversityHospital of Sichuan University, Chengdu, Sichuan
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Tianjin Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No